CLINICAL TRIAL: NCT02948907
Title: Endobronchial Ultrasound "Elastography" and "Tissue Harmonic Imaging" for Characterisation of Hilar and Mediastinal Lymph Nodes
Brief Title: "Elastography" and "Tissue Harmonic Imaging" for Characterisation of Hilar and Mediastinal Lymph Nodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Prof. Dr. med., Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Protocol F1.0 - 22/05/2013
Record Dates: First submitted 2016-09-19; First posted 2016-10-31 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Lymphadenopathy
MeSH Terms: conditions — Lymphadenopathy | interventions — Bronchoscopy

ARMS (1):
- Procedure/Bronchoscopy (Other): Patients with enlarged hilar and/or mediastinal lymph nodes and indication for EBUS-TBNA undergo diagnostic bronchoscopy. For characterisation of the enlarged lymph nodes, endobronchial ultrasound with elastography and "Tissue Harmonic Imaging (THI)" are used. Afterwards, EBUS-TBNA is performed. The results of elastography and THI are correlated with the cytological results obtained by EBUS-TBNA.
  Interventions: Other: Procedure/Bronchoscopy

INTERVENTIONS:
Other: Procedure/Bronchoscopy — Patients with enlarged hilar and/or mediastinal lymph nodes and indication for EBUS-TBNA undergo diagnostic bronchoscopy. For characterisation of the enlarged lymph nodes endobronchial ultrasound with elastography and "Tissue Harmonic Imaging (THI)" are used. Afterwards, EBUS-TBNA is performed. The results of elastography and THI are correlated with the cytological result obtained by EBUS-TBNA.

SUMMARY:
Several benign and malignant diseases are associated with hilar and mediastinal lymphadenopathy. Endobronchial elastography that is an imaging procedure used for the visualization of tissue elasticity and "Tissue Harmonic Imaging (THI)" might be useful for the differentiation of benign and malignant lymph nodes.

DETAILED DESCRIPTION:
Patient enrolment and data acquisition is to be carried out on a prospective basis. Patients with hilar and/or mediastinal lymphadenopathy and indication for EBUS-TBNA are enroled. It is planned to evaluate 100 lymph nodes by elastography and THI. All patients will undergo diagnostic bronchoscopy at one study centre in Heidelberg.

ELIGIBILITY:
Inclusion Criteria:

* Indication for EBUS-TBNA
* Patient has provided written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-12-01 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of elastography and "Tissue Harmonic Imaging" | Once after bronchoscopic procedure
  Correlation of imaging results and cytological results after bronchoscopic procedure

SECONDARY OUTCOMES:
Safety of endobronchial use of elastography and "Tissue Harmonic Imaging" assessed by Incidence of adverse events | during diagnostic bronchoscopy procedure
  Incidence of adverse events (e.g. bleeding, pneumothorax)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD, Principal Investigator — Thoraxklinik at University of Heidelberg
Locations (1):
- Thoraxklinik, Heidelberg, Germany

REFERENCES:
- [Result] Gompelmann D, Kontogianni K, Sarmand N, Kaukel P, Krisam J, Eberhardt R, Herth FJF. Endobronchial Ultrasound Elastography for Differentiating Benign and Malignant Lymph Nodes. Respiration. 2020;99(9):779-783. doi: 10.1159/000509297. Epub 2020 Oct 7. PMID 33027791